CLINICAL TRIAL: NCT05992207
Title: Motor Imagery Training for Improvement of Balance of Ataxic Children
Brief Title: Utilization of Motor Imagery Training for Improvement of Balance of Ataxic Children After Medulloblastoma Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Saeed Alsakhawi, Assisstant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/ 012/004454
Record Dates: First submitted 2023-07-19; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Cerebellar Ataxia
MeSH Terms: conditions — Cerebellar Ataxia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical thertapy training (Active Comparator): The Control group received the selected physical therapy program for one hour, three times weekly for three successive months including facilitation of balance and protective reactions from standing position, standing on one leg, weight shifting from standing, squat to standing, strengthening exercises for trunk muscles and for upper and lower extremities musculatures, gait training activities for correction of gait pattern
  Interventions: Other: physical therapy training
- motor imaginary training (Active Comparator): The study group received the selected physical therapy program for one hour, three times weekly for three successive months in addition to motor imagery program for 30 minutes as the following. Each child shown a video of 5 minutes of illustrating normal movements while the child resting in semireclined sitting in quiet room in front the screen. Children then asked to close their eyes and imagine practicing the task like the illustrative video. Repetition of the exercises depend on the children ranging from 5 to 10 repetitions per exercise
  Interventions: Other: motor imaginary training

INTERVENTIONS:
Other: motor imaginary training — Each child shown a video of 5 minutes of illustrating normal movements while the child resting in semi#reclined sitting in quiet room in front the screen. Children then asked to close their eyes and imagine practicing the task like the illustrative video. Repetition of the exercises depend on the children ranging from 5 to 10 repetitions per exercise.
  Arms: motor imaginary training
Other: physical therapy training — facilitation of balance and protective reactions from standing position, standing on one leg, weight shifting from standing, squat to standing, strengthening exercises for trunk muscles and for upper and lower extremities musculatures, gait training activities for correction of gait pattern
  Arms: physical thertapy training

SUMMARY:
Background: after resection of medulloblastoma in children they suffer from signs and symptoms of ataxia which impedes their activities of daily living. purpose: to investigate the effect motor imagery training on balance, severity of ataxia and gait parameters on children after resection of medulloblastoma. Methods: Fifty children surfing from cerebellar ataxia after medulloblastoma resection were selected from tumors hospital of Cairo University, their age ranged from seven to nine years old, they were randomly assigned into two matched control and study groups. The control groups received the selected physical therapy program while, the study group received motor imaginary training in addition to the selected physical therapy program. Both groups were evaluated by ataxic rating scale, pediatric berg balance scale and kinematic gait analysis by kinovea software.

DETAILED DESCRIPTION:
Motor imagery is an effective method to enhance motor performance applied in rehabilitation programs it did not impose a physical load on patients, was confirmed through clinical evidence from meta#analysis. Motor imagery means thinking in motor task with executing it to activate motor cortical areas as 25% of the brain neurons are mirror neurons and fire by thinking.

ELIGIBILITY:
Inclusion Criteria:

* The children had signs of ataxia
* loss of balance
* able to understand and execute test instructions
* the children are in the follow up period after medulloblastoma resection

Exclusion Criteria:

* medically unstable
* visual impairment
* increased intracranial pressure
* any other neuromuscular diseases.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-01-21 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Severity of ataxia | 3 months
  The SARA determines the degree of ataxia. It has eight items with a score range of 0 (means no ataxia) to 40 (means severe ataxia). It contains sitting, stance, gait, limb kinetic functions, heel-shin slide, fast alternating hand movements, nose-finger test, finger chase, and speech disturbance. The arithmetic means of the left and right sides and independent ratings of each side are included in the SARA total score.
Pediatric berg balance scale | 3 months
  The Paediatric Berg Balance Scale assesses children's balance. The scale includes 14 items: sit to stand, stand to sit, transfers, stand unsupported, sit unsupported, stand with eyes closed, stand with feet together, stand with one foot in front of the other, stand on one foot, turn 360 degrees, turn to look behind, retrieve an object from the floor, place an alternating foot on a stool, and reach forward with an outstretched arm. The total scale score ranges from zero to 56.
Kinematic gait assessment | 3 months
  Kinematic gait analysis measured temporospatial gait variables using a two-dimensional motion analysis system. Markers were placed on the skin overlying the lateral femoral epicondyle, greater trochanter, 5th metatarsal head, and lateral malleolus. The therapist set a tripod with a fixed video camera at 3 m from the walkway. The fixed video camera was concentrated on the central part to record three gait cycles in the sagittal plane. The therapist used the Kinovea software (version 8.15.0) to measure stride length, step length, cadence, and walking speed. The measurement involved one walking trial at the chosen speed throughout the 4-m walkway.

CONTACTS AND LOCATIONS:
Overall Officials: Reham Alsakhawi, Principal Investigator — Cairo University
Locations (1):
- Reham Alsakhawi, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data from participants will be made available
Supporting Information: Study Protocol
Time Frame: 12 months after study completion
Access Criteria: data access requests will be reviewed by an external independent review panel. requestor will be required to sign a data access agreement

REFERENCES:
- [Derived] Alsakhawi RS, Elshafey MA, Alkhouli MN. Utilization of Motor Imagery Training for Improvement of Balance of Ataxic Children after Medulloblastoma Resection. Sci Rep. 2024 Nov 27;14(1):29500. doi: 10.1038/s41598-024-78900-7. PMID 39604382